CLINICAL TRIAL: NCT02032927
Title: A COMPARATIVE STUDY BETWEEN TWO PHARMACOLOGICAL ASSOCIATIONS OXYCODONE/NALOXONE AND CODEINE / PARACETAMOL IN TREATMENT OF MODERATE-SEVERE CHRONIC PAIN DUE TO OSTEOARTHRITIS OF KNEE AND/OR HIP
Brief Title: Treatment of Chronic Pain From Osteoarthritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-SM-14-OA
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain
Keywords: osteoarthritis; pain; opioids
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Pain | interventions — acetaminophen, codeine drug combination; Oxycodone; Naloxone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Codeine/paracetamol (Active Comparator): The combination codeine/paracetamol,30 mg/500 mg,1 tablet every 8 hours, paracetamol 500 mg if NRS> 4, repeatable up to 3 times per day.
  At any stage of the study, patients treated with combination codeine/paracetamol in case of ineffectiveness (NRS> 4) despite maximal dosage (2 tablets every 8 hours) and/or side effect, will be subject to the opioid switch and will start equianalgesic therapy with oxycodone/naloxone combination.
  Interventions: Drug: Codeine/paracetamol
- Oxycodone/Naloxone (Active Comparator): Combination oxycodone /naloxone, 5 mg/2.5 mg, 1 tablet/day, paracetamol 500 mg if NRS> 4, repeatable up to 3 times per day.
  Interventions: Drug: Oxycodone/naloxone

INTERVENTIONS:
Drug: Codeine/paracetamol — Randomization to one of the two treatments will be done through appropriate randomization list.
  During the first 15 days of treatment in the event of failure of efficacy, understood as the average pain intensity higher than 4 (monitored with NRS) with the need to take more than two rescue doses of paracetamol per day, and in the absence of side effects, the patients will be instructed on how to proceed with dosage adjustments according to specific guidelines.
  The patient will be evaluated at 15 days, 1 month, 2 months and three months. Your health care professional who administer the assessment scales (WOMAC, SF-12, BFI, TMT) will not know in any way which treatment the patient is taking.
  Arms: Codeine/paracetamol
Drug: Oxycodone/naloxone — Randomization to one of the two treatments will be done through appropriate randomization list.
  During the first 15 days of treatment in the event of failure of efficacy, understood as the average pain intensity higher than 4 (monitored with NRS) with the need to take more than two rescue doses of paracetamol per day, and in the absence of side effects, the patients will be instructed on how to proceed with dosage adjustments according to specific guidelines.
  The patient will be evaluated at 15 days, 1 month, 2 months and three months. Your health care professional who administer the assessment scales (WOMAC, SF-12, BFI, TMT) will not know in any way which treatment the patient is taking.
  Arms: Oxycodone/Naloxone

SUMMARY:
Osteoarthritis is a common joint disorder in the elder population.The current treatment options include both a non-pharmacological approach (physiokinesitherapy, diet) or if this fails, a pharmacological approach that relies in the first instance on drugs such as paracetamol, non-steroidal anti-inflammatory (including inhibitors of cyclo-oxygenase). However, the use of these drugs is limited, by the roof effect concerning analgesia, and by the potential side effects. When pharmacological treatments with non-opioid medications fail, and a moderate-to-severe pain reduces the quality of life of the patient, international guidelines suggest the use of opioid drugs.

DETAILED DESCRIPTION:
The WHO analgesic ladder, even with its limitations, is widely used to guide the beginning of opioid therapy in chronic pain. According to this approach the choice of drug is based on the intensity of pain reported by the patient; belong to the first step acetaminophen and nonsteroidal anti-inflammatory drugs (NSAIDs), and if these drugs fail it is planned to introduce a weak opioid (tramadol, codeine) alone or in combination.

The association codeine-paracetamol, one of the most widely used drug combinations in the treatment of moderate pain from osteoarthritis, demonstrated analgesic efficacy superior only to paracetamol in the short term; however, its use was less effective in the long term and worsen by multiple side effects, especially gastrointestinal with results in poor adherence to the therapy.

Lately, the international guidelines on the treatment of chronic pain in cancer have suggested the possibility of moving, in case of inadequate efficacy of paracetamol and / or NSAIDs, directly to the third step, using a low dose of a strong opioid.

The side effects associated with the use of opioids in the treatment of chronic pain, such as itching, side effects of gastrointestinal and central nervous system effects (drowsiness, giddiness), often necessitate dose reduction (thus compromising the analgesic effect), with often resulting in discontinuation of treatment.

A recent strategy to face the underlying cause of opioid-induced constipation (OIC) is the oral administration of an antagonist of opioid receptor that acts specifically and locally at the level of the gastrointestinal tract. This prevents or minimizes gastrointestinal side effects but does not affect the central analgesic effect of the opioid thank to the low bioavailability of the antagonist.

A recent review on the effects of chronic pain on cognitive function of patients describes a series of clinical evidence suggestive of a intellectual impairment predominantly associated with a significant psychomotor slowing.

An interesting corollary of the problematic pain-cognition is represented by the possible neuropsychological side effect due to teh use of opioid drugs in the treatment of chronic pain.

The objective of the research becomes to determinate how much the analgesic relief, derived from the assumption of opioid drugs, can lead to an improvement in cognitive function without the possible side effects of the drugs themselves.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 60 years old
* Individuals with a primary diagnosis of osteoarthritis
* Subject that are able to understand the purpose of the study and that have signed a written informed consent
* Subjects that are able to take prescribed therapies, understand and complete the questionnaires and forms

Exclusion Criteria:

* Subject with history of hypersensitivity to oxycodone, naloxone , codeine , acetaminophen, ibuprofen, and the other ingredients in the formulations studied
* Subjects with known structural alterations in the gastrointestinal tract
* Subjects with secondary osteoarthritis
* Subjects with history of abuse of alcohol and / or drugs
* Subjects with history of abuse opioids.
* Patients suffering from rheumatoid arthritis
* Patients with evidence of medical or surgical unstable
* Patients with current or previous history of epilepsy
* Patients treated with anti-depressive action on the central nervous system which in the opinion of the investigator may result in additive effects with the drugs under study.
* Subjects with renal and / or hepatic impairment severe
* Subjects with a history of depression or other psychiatric condition that, in the opinion of the investigator might interfere with the study participation
* Individuals with cognitive impairment

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluate differences in terms of efficacy and tolerability between two pharmaceutical protocols in patients with chronic pain due to osteoarthritis. | 15 days from the enrolment
  The number of patients has been estimated considering that, at 15 days of enrollment, a reduction of 30% of the WOMAC pain subscale, with a score at BFI <50, the use of not more than one laxative drug or the absence of side effects such as to consider the need to discontinue therapy occurs in 80% of patients in Protocol B versus 50% of patients in Protocol A, with 73 patients per group will be able to highlight an odds ratio (OR) 2.65 with a power of 80% and an alpha error of 5% (2-tailed). The calculation was performed with nQuery 4 (Statistical Solutions, Cork, IRL).
  Considering a drop out rate of about 24% is numerosity you plan to enroll a total of 182 patients in order to obtain 146 patients valid.

SECONDARY OUTCOMES:
Evaluate the differences between the two drug protocols, in terms of quality of life, by using of the SF-12 questionnaire. | 3 months from the enrollment
Evaluation of the differences between the two drug protocols, in the scores obtained in the two sections, functionality and rigidity of the WOMAC questionnaire. | 3 months from the enrollment
The evaluation of the attentive functions (selective and divided attention) and of eye-manual coordination and of psycho-motor speed will be performed trough Trail Making Test (Reitan, 1944) to all patients enrolled for the project. | 3 months from the enrollment
  The secondary endpoints, all on a continuous scale, will be analyzed using the Mann-Whitney U test; for each group will be reported median and quartiles.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Principal Investigator — IRCCS Fondazione San Matteo Pavia
Locations (14):
- Italy (14):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - Azienda Ospedaliera della Provincia di Pavia - Ospedale "Carlo Mira" - U.O. Medicina Interna - Servizio di Anestesia e Rianimazione - Ambulatorio di Terapia del dolore, Casorate Primo
  - Azienda Istituti Ospitalieri di Cremona, Presidio Ospedaliero di Cremona - U.O. di Anestesia, Analgesia e Medicina Perioperatoria, Cremona
  - Azienda Ospedaliera della provincia di Lodi Dipartimento emergenza urgenza, Lodi
  - Azienda Ospedaliera Istituto Ortopedico Gaetano Pini - U.O.C. Anestesia e Rianimazione, Milan
  - Azienda Ospedaliera della Provincia di Pavia - Ospedale Asilo Vittoria di Mortara - U.O. di Pneumotisiologia, Mortara
  - Clinica San Carlo - Casa di Cura Polispecialistica S.p.A. - Unità di Terapia del Dolore, Paderno Dugnano
  - Azienda Servizi alla Persona, ASP, "II.AA.RR." - Istituto di Riabilitazione "Santa Margherita" - Struttura Complessa di Riabilitazione, Pavia
  - Fondazione Salvatore Maugeri - sede di Via Boezio - UO Cure Palliative e Terapia del Dolore, Pavia
  - IRCCS Istituto Clinico "Humanitas" - Anestesia, Day Hospital chirurgico - Chronic Pain Service, Rozzano
  - Dipartimento Integrato di Lungassistenza Anziani - ASL TO1, Torino
  - Ospedale di circolo Fondazione Macchi - SSD Anestesia Day Surgery, Varese
  - Azienda Ospedaliera della Provincia di Pavia - Ospedale Civile di Vigevano - Servizio di Anestesia e Rianimazione, Vigevano
  - Azienda Ospedaliera della Provincia di Pavia - Ospedale Civile di Voghera- U.O. di Medicina Interna - U.O. di Riabilitazione specialistica, Voghera